CLINICAL TRIAL: NCT06945978
Title: Validation of a miRNA Panel to Optimize Treatment Response in Patients With Metastatic Pancreatic Cancer
Brief Title: Validation of a miRNA Panel to Optimize Treatment Response in Patients With Metastatic Pancreatic Cancer (mirPANC 2)
Acronym: mirPANC 2
Status: Recruiting | Type: Observational
Sponsor: Benedito Mauro Rossi (Other)
Responsible Party: Sponsor-Investigator, Benedito Mauro Rossi, Surgeon Oncologist, Beneficência Portuguesa de São Paulo
Organization: Beneficência Portuguesa de São Paulo (Other)
Other Study IDs: mirPANC 2
Record Dates: First submitted 2025-03-18; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer; Metastasis; Epigenetic
Keywords: Pancreatic cancer; miRNA; Treatment response; Epigenetic; Folfirinox
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — miRNA, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-responder: Patients who do not respond to the FOLFIRINOX regimen.
- Responder: Patients who respond to the FOLFIRINOX regimen.

SUMMARY:
This study is being conducted to better understand how pancreatic cancer behaves during treatment and how we can improve methods for monitoring disease progression. The research aims to determine whether small molecules present in the blood, called miRNAs, can help doctors assess whether the treatment is working or needs adjustment. With this, we hope to make cancer monitoring less invasive and more precise, allowing patients to receive more personalized and effective treatments.

DETAILED DESCRIPTION:
Pancreatic cancer, particularly Pancreatic Ductal Adenocarcinoma (PDAC), has an extremely poor prognosis, with a 5-year survival rate of less than 3% for advanced stages. In 2020, Brazil saw about 11,893 deaths from this condition, with incidence rates expected to rise. The standard treatment for metastatic PDAC is the FOLFIRINOX regimen, but its response is variable and its effectiveness is limited, with few advancements in personalized therapy and response prediction. This research aims to develop and validate a panel of serum-based miRNA biomarkers using qPCR and large-scale sequencing (NGS) to evaluate treatment response in metastatic PDAC patients. The goal is to identify miRNA expression patterns that predict the effectiveness of FOLFIRINOX and assist in personalizing treatment based on individual responses. The study will use liquid biopsy to collect blood samples and analyze circulating miRNAs, enabling early detection of treatment responses and disease progression. This will allow for precise therapeutic adjustments and alternative treatment options based on the patient's profile. The innovative approach combines liquid biopsy with miRNA analysis as a low-cost, effective tool for monitoring and personalizing treatment. Using qPCR, a more affordable method than NGS and microarrays, enhances clinical feasibility. The research is highly relevant to the Brazilian Unified Health System (SUS), as an accessible miRNA panel could optimize resource use, reduce costs of ineffective treatments, and improve care quality and outcomes, aligning with SUS's goals for precise and accessible healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic PDAC;
* Patients who will start treatment with FOLFIRINOX;
* 18 years or older;
* Who agree to participate in the study by signing the Informed Consent Form;

Exclusion Criteria:

* Patients who have previously undergone chemotherapy, whether neoadjuvant, adjuvant, or any prior first-line treatment;
* Patients who do not meet the minimum criteria to receive the proposed regimen, such as those with hyperbilirubinemia, those who are not candidates due to age or performance status deterioration;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with metastatic PDAC of both sexes, aged 18 years or older, who will start treatment with FOLFIRINOX at BP - A Beneficência Portuguesa de São Paulo.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | After 4 cycle of therapy (each cycle is 15 days)
  Response to FOLFIRINOX treatment after 4 cycles of therapy.
Response to treatment | After the 8 cycle of therapy (each cycle is 15 days)
  Response to FOLFIRINOX treatment after 8 cycles of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- A Beneficência Portuguesa de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No